CLINICAL TRIAL: NCT06740136
Title: Genetic Determinants of Exercise-Induced Muscle Damage (POLYGENDOMUS) / Déterminants Génétiques Des Dommages Musculaires Induits Par L'exercice (POLYGENDOMUS)
Brief Title: Genetic Determinants of Exercise-Induced Muscle Damage (POLYGENDOMUS)
Acronym: POLYGENDOMUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-007; 2022-A01308-35 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-12-10; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Muscle damage; Single nucleotide polymorphism; exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Intervention model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): exercise group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Muscle induced-damage eccentric exercise

SUMMARY:
The objective of this study is to evaluate the association between the evolution of plasma CPK levels and genetic polymorphisms, both before the muscle-damaging exercise and at three post-exercise time points. The investigators aim to include 300 participants in this research.

DETAILED DESCRIPTION:
Elite-level sports expose athletes to training loads designed to induce muscle damage, aiming to achieve optimal physiological adaptations. However, the repetitive nature of such damage increases the risk of injury. The ability to assess an athlete's susceptibility to fragility is therefore crucial for optimizing their training and performance. Genetic factors appear to play a significant role in the occurrence of these injuries, particularly through subtle variations in DNA sequences. Depending on the location of these variations within a gene, they may or may not alter the expression or function of the associated protein. The investigators aimed to investigate the relationship between genetic polymorphisms and biological parameters in the context of exercise-induced muscle damage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between 18 and 35
* Weighing more than 50 kg
* Member of a sports club affiliated to an Olympic federation
* Socially insured
* Willing to comply with all study procedures and duration of the study

Exclusion Criteria:

* Medical history contraindicating sporting activities
* Current medical treatment
* Not a member of a sports club affiliated to an Olympic federation
* Administrative reasons: impossibility of receiving informed information, impossibility of participating in the entire study, absence of social security coverage, refusal to sign consent form.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
The association between single nucleotide polymorphisms and exercise induced blood creatine kinase variation | Evolution of kinetics from Day 0 to Day 3 post experiment
  Association between blood creatine kinase level variations and single nucleotide polymorphisms.
  The Outcome Measure in this study is focused on the variation in plasma CPK levels following an exercise inducing muscle damage. The result is expressed as a change in plasma CPK concentration, measured in units per liter (U/L). This single measurement is used to investigate its association with genetic polymorphisms. Therefore a regression analysis will be performed to identify the association. This study is exploratory and the genetic polymorphisms are not pre-identified but will be investigated through a comprehensive analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasport, Loos, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://urepsss.univ-lille.fr/